CLINICAL TRIAL: NCT00835770
Title: A Dose-Blind, Multicenter, Extension Study to Determine the Long-Term Safety and Efficacy of Two Doses of BG00012 Monotherapy in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: BG00012 Monotherapy Safety and Efficacy Extension Study in Multiple Sclerosis (MS)
Acronym: ENDORSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS303; 2008-004753-14 (EudraCT Number)
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: relapsing; multiple sclerosis; remitting; oral
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Recurrence; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG00012 plus placebo (Experimental): In the first phase, participants will receive BG00012 240 mg (two 120 mg capsules) twice a day (BID) and 2 placebo capsules once a day. In the second phase participants will receive open-label BG00012 240 mg BID, for atleast 8 years.
  Interventions: Drug: dimethyl fumarate; Drug: Placebo
- BG00012 (Experimental): In the first phase participants will receive BG00012 240 mg (two 120 mg capsules) three times a day (TID). In the second phase participants will receive open-label BG00012 240 mg BID for atleast 8 years.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — BG00012 capsules
  Other Names: BG00012; Tecfidera; DMF
Drug: Placebo — Capsules taken to maintain the blind in the 240 mg BID treatment group.
  Arms: BG00012 plus placebo

SUMMARY:
The primary objective of this study is to evaluate the long-term safety profile of BG00012 (dimethyl fumarate). Secondary objectives of this study are to evaluate the long-term efficacy of BG00012 using clinical endpoints and disability progression, to evaluate further the long-term effects of BG00012 on multiple sclerosis (MS) brain lesions on magnetic resonance imaging (MRI) scans in participants who had MRI scans as part of Studies 109MS301 (NCT00420212) and 109MS302 (NCT00451451) and to evaluate the long-term effects of BG00012 on health economics assessments and the visual function test.

DETAILED DESCRIPTION:
The initial BG00012 dosage for the extension study (240 mg BID or 240 mg TID) was the same as that used in the Phase 3 Studies 109MS301 (NCT00420212) and 109MS302 (NCT00451451). Subsequent to the initiation of this study, BG00012 was approved in several countries for the treatment of MS at a dose of 240 mg BID. For this reason, all participants continuing in this study will receive the currently marketed dose of 240 mg BID.

ELIGIBILITY:
Key Inclusion Criteria:

-Subjects who participated in and completed as per protocol previous BG00012 clinical studies 109MS301 (NCT00420212) or 109MS302 (NCT00451451).

Key Exclusion Criteria:

* Any significant change in medical history from 109MS301 or 109MS302 that would have excluded subject's participation from their previous study.
* Subjects from 109MS301 or 109MS302 who discontinued oral study treatment due to an AE or due to reasons other than protocol-defined relapse/disability progression.
* Subjects from 109MS301 or 109MS302 who discontinued study treatment due to disability progression or relapses and did not follow the modified visit schedule up to Week 96.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 19 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1736 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (204):
- United States (47):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Loma Linda, California
  - Research Site, Boulder, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, North Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Albany, New York
  - Research Site, Amherst, New York
  - Research Site, Buffalo, New York
  - Research Site, Patchogue, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Bellevue, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Rumford, Rhode Island
  - Research Site, Cordova, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Issaquah, Washington
  - Research Site, Madison, Wisconsin
- Australia (8):
  - Research Site, Kogarah, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Melbourne, Victoria
  - Research Site, Box Hill
  - Research Site, Chatswood
  - Research Site, Fitzroy
  - Research Site, Geelong
  - Research Site, Sydney
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Belarus (3):
  - Research Site, Belarus, Homyel’ Voblasc’
  - Research Site, Belarus’, Vitebsk Oblast
  - Research Site, Minsk
- Belgium (10):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Damme
  - Research Site, Diepenbeek
  - Research Site, Hechtel-Eksel
  - Research Site, Leuven
  - Research Site, Lodelinsart
  - Research Site, Sint-Truiden
- Research Site, Tuzla, Bosnia and Herzegovina
- Bulgaria (2):
  - Research Site, Rousse
  - Research Site, Sofia
- Canada (7):
  - Research Site, Lévis, Quebec
  - Research Site, Edmonton
  - Research Site, London
  - Research Site, Montreal
  - Research Site, Nova Scotia
  - Research Site, Ottawa
  - Research Site, Regina
- Research Site, Zagreb, Croatia
- Czechia (8):
  - Research Site, Brno
  - Research Site, Jihlava
  - Research Site, Moravská Ostrava
  - Research Site, Olomouc
  - Research Site, Opava
  - Research Site, Ostrava - Vítkovice
  - Research Site, Prague
  - Research Site, Teplice
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (13):
  - Research Site, Amiens
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
- Germany (23):
  - Research Site, Berg, Bavaria
  - Research Site, Steinfurt, Ibbenbueren
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Erbach im Odenwald
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, Minden
  - Research Site, Munich (München)
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Regensburg
  - Research Site, Westerstede
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chandigarh
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Ludhiana
  - Research Site, Mangalore
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
- Research Site, Dublin, Ireland
- Israel (3):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Safed
- Research Site, Roma, Italy
- Research Site, Riga, Latvia
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Morelia
  - Research Site, San Luis Potosí City
- Research Site, Chisinau, Moldova
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Geleen
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Hamilton
- Research Site, Skopje, North Macedonia
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lódz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Plewiska
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Guaynabo, Puerto Rico
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Târgu Mures
  - Research Site, Timișoara
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Martin
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Durban
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Ukraine (8):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (5):
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Amezcua L, Mao-Draayer Y, Vargas WS, Farber R, Schaefer S, Branco F, England SM, Belviso N, Lewin JB, Mendoza JP, Shankar SL; ENDORSE Study Investigators. Efficacy of Dimethyl Fumarate in Young Adults with Relapsing-Remitting Multiple Sclerosis: Analysis of the DEFINE, CONFIRM, and ENDORSE Studies. Neurol Ther. 2023 Jun;12(3):883-897. doi: 10.1007/s40120-023-00475-8. Epub 2023 Apr 15. PMID 37061656
- [Derived] Gold R, Arnold DL, Bar-Or A, Fox RJ, Kappos L, Chen C, Parks B, Miller C. Safety and efficacy of delayed-release dimethyl fumarate in patients with relapsing-remitting multiple sclerosis: 9 years' follow-up of DEFINE, CONFIRM, and ENDORSE. Ther Adv Neurol Disord. 2020 May 12;13:1756286420915005. doi: 10.1177/1756286420915005. eCollection 2020. PMID 32426039
- [Derived] Mehta D, Miller C, Arnold DL, Bame E, Bar-Or A, Gold R, Hanna J, Kappos L, Liu S, Matta A, Phillips JT, Robertson D, von Hehn CA, Campbell J, Spach K, Yang L, Fox RJ. Effect of dimethyl fumarate on lymphocytes in RRMS: Implications for clinical practice. Neurology. 2019 Apr 9;92(15):e1724-e1738. doi: 10.1212/WNL.0000000000007262. Epub 2019 Mar 27. PMID 30918100
- [Derived] Gold R, Giovannoni G, Phillips JT, Fox RJ, Zhang A, Marantz JL. Sustained Effect of Delayed-Release Dimethyl Fumarate in Newly Diagnosed Patients with Relapsing-Remitting Multiple Sclerosis: 6-Year Interim Results From an Extension of the DEFINE and CONFIRM Studies. Neurol Ther. 2016 Jun;5(1):45-57. doi: 10.1007/s40120-016-0042-8. Epub 2016 Mar 1. PMID 26932146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 298 investigative sites from 03 February 2009 to 08 November 2019.
Pre-assignment Details: The study included participants who completed studies NCT00420212 and NCT00451451. A total of 1736 participants were treated in the open label phase extension study NCT00835770, out of which 759 completed the study.
Groups:
- BG00012 240 mg BID: Participants received BG00012 240 milligram (mg), 2 capsules (120 mg each) orally, twice a day (BID) and 2 matching placebo capsules once a day (QD) for up to 8 years.
- BG00012 240 mg TID: Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, three times a day (TID) for up to 8 years.
Period: Overall Study
Arm/Group | BG00012 240 mg BID | BG00012 240 mg TID
Started | 868 | 868
Completed | 384 | 375
Not Completed | 484 | 493
Not completed — MS Relapse | 17 | 23
Not completed — MS Progression | 14 | 9
Not completed — Adverse Event | 113 | 124
Not completed — Lost to Follow-up | 22 | 19
Not completed — Consent Withdrawn | 144 | 156
Not completed — Investigator Decision | 42 | 42
Not completed — Participant Non-Compliance | 11 | 9
Not completed — Death | 4 | 6
Not completed — Other | 115 | 104
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included participants who had entered study NCT00835770 and received at least one dose of study treatment. Data for ethnicity was not evaluated in the study.
Groups:
- BG00012 240 mg BID: Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, BID and 2 matching placebo capsules QD for up to 8 years.
- BG00012 240 mg TID: Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, TID for up to 8 years.
- Total: Total of all reporting groups
Arm/Group | BG00012 240 mg BID | BG00012 240 mg TID | Total
Number analyzed (Participants) | 868 | 868 | 1736
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (8.93) | 40.1 (9.23) | 39.8 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 616 | 596 | 1212
  Male | 252 | 272 | 524
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 285 | 309 | 594
  Black or African American | 10 | 16 | 26
  Asian | 82 | 80 | 162
  Other | 32 | 24 | 56
  Not Reported Due To Confidentiality Regulations | 459 | 439 | 898

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Day 1 up to Week 561
Population: Safety population included all participants who had any post-baseline safety follow-up in study NCT00835770, defined as any treatment emergent AE in study NCT00835770 or any post-baseline laboratory, vital signs, or physical exam assessment in study NCT00835770, and received at least one dose of study treatment in study NCT00835770.
Measure: Count of Participants; unit: Participants
Arm/Group | BG00012 240 mg BID | BG00012 240 mg TID
Number analyzed (Participants) | 868 | 868
Participants | 824 | 814

2. Secondary Outcome: Percentage of Participants Who Had Relapses
Description: Relapses were defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours.
Time Frame: Day 1 up to Week 384
Population: ITT population included participants who had entered study NCT00835770 and received at least one dose of study treatment. Data for this outcome measure (OM) was summarized as per treatment received in previous studies (NCT00420212 and NCT00451451).
Measure: Number; unit: percentage of participants
Groups:
- BG00012 240 mg BID (Prior BG00012 240 mg BID): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, BID and 2 matching placebo capsules QD for up to 8 years. Participants who had received BG00012 240 mg BID in the previous studies were included in this arm group.
- BG00012 240 mg TID (Prior BG00012 240 mg TID): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, TID for up to 8 years. Participants who had received BG00012 240 mg TID in the previous studies were included in this arm group.
- BG00012 240 mg BID (Prior BG00012 Matched Placebo): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, BID and 2 matching placebo capsules QD for up to 8 years. Participants who had received placebo matched to BG00012 in the previous studies were included in this arm group.
- BG00012 240 mg TID (Prior BG00012 Matched Placebo): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, TID for up to 8 years. Participants who had received placebo matched to BG00012 in the previous studies were included in this arm group.
- BG00012 240 mg BID (Prior Glatiramer Acetate [GA]): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, BID and 2 matching placebo capsules QD for up to 8 years. Participants who had received Glatiramer Acetate (GA) in the previous studies were included in this arm group.
- BG00012 240 mg TID (Prior Glatiramer Acetate [GA]): Participants received BG00012 240 mg, 2 capsules (120 mg each) orally, TID for up to 8 years. Participants who had received GA in the previous studies were included in this arm group.
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
percentage of participants | 40 | 41 | 34 | 36 | 31 | 31

3. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: The annualized relapse rate is calculated as the total number of relapses occurred during the period for all participants, divided by the total number of participant-years followed in the period.
Time Frame: Day 1 up to Week 384
Population: ITT population included participants who had entered study NCT00835770 and received at least one dose of study treatment. Data for this OM was summarized as per treatment received in previous studies (NCT00420212 and NCT00451451).
Measure: Number; unit: relapses per participant-years
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
relapses per participant-years | 0.159 | 0.179 | 0.200 | 0.199 | 0.184 | 0.212

4. Secondary Outcome: Change From Baseline in the Expanded Disability Status Scale (EDSS) at Week 384
Description: EDSS scale ranges from 0 (Normal neurological exam, no disability) to 10 (Death) in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. Sustained disability progression was defined as at least a 1.0 point increase on the EDSS from a baseline EDSS ≥1.0 that was sustained for at least 24 weeks, or a 1.5 point increase on the EDSS from a baseline EDSS =0 that was sustained for at least 24 weeks.
Time Frame: Baseline, Week 384
Population: ITT population included participants who had entered study NCT00835770 and received at least one dose of study treatment. 'Number Analyzed' =Number of participants analyzed at specific timepoint. Data for this OM was summarized as per treatment received in previous studies (NCT00420212 and NCT00451451).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
score on a scale
  Baseline: number analyzed (Participants) | 499 | 502 | 249 | 248 | 118 | 118
  Baseline | 2.44 (1.251) | 2.43 (1.144) | 2.50 (1.135) | 2.54 (1.218) | 2.57 (1.249) | 2.68 (1.231)
  Change at Week 384: number analyzed (Participants) | 226 | 219 | 90 | 98 | 42 | 50
  Change at Week 384 | 0.28 (1.160) | 0.26 (1.213) | 0.37 (1.328) | 0.53 (1.278) | 0.39 (1.217) | 0.49 (1.319)

5. Secondary Outcome: Number of Gadolinium (Gd)-Enhancing Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The Gd-enhancing lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: MRI population. 'Number Analyzed' =Number of participants analyzed at specific timepoint. Data for this OM was summarized as per treatment received in previous studies (NCT00420212 and NCT00451451).
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
lesions
  Week 48: number analyzed (Participants) | 191 | 195 | 83 | 78 | 41 | 48
  Week 48 | 0.4 (1.87) | 0.4 (1.29) | 0.2 (0.66) | 0.3 (1.14) | 0.5 (1.19) | 0.4 (1.14)
  Week 96: number analyzed (Participants) | 183 | 186 | 77 | 75 | 39 | 46
  Week 96 | 0.4 (1.77) | 0.4 (1.28) | 0.1 (0.38) | 0.2 (0.82) | 0.6 (1.33) | 0.3 (0.73)
  Week 144: number analyzed (Participants) | 156 | 159 | 66 | 60 | 32 | 41
  Week 144 | 0.3 (1.66) | 0.4 (1.30) | 0.2 (0.44) | 0.1 (0.29) | 0.5 (2.48) | 0.3 (1.59)
  Week 192: number analyzed (Participants) | 144 | 149 | 59 | 55 | 33 | 38
  Week 192 | 0.4 (2.02) | 0.5 (1.85) | 0.5 (1.72) | 0.3 (0.96) | 0.2 (0.60) | 0.6 (2.01)
  Week 240: number analyzed (Participants) | 135 | 134 | 55 | 53 | 29 | 34
  Week 240 | 0.5 (3.14) | 0.5 (2.29) | 0.2 (0.50) | 0.2 (0.51) | 0.2 (0.58) | 0.3 (0.75)
  Week 288: number analyzed (Participants) | 90 | 97 | 30 | 32 | 6 | 16
  Week 288 | 0.2 (0.74) | 0.5 (1.81) | 0.1 (0.40) | 0.7 (2.76) | 0.0 (0.00) | 0.3 (0.77)

6. Secondary Outcome: Volume of Gd-Enhancing Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The Gd-enhancing lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter cube (mm^3)
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
millimeter cube (mm^3)
  Baseline: number analyzed (Participants) | 209 | 220 | 104 | 99 | 47 | 60
  Baseline | 31.7 (179.28) | 48.6 (205.43) | 96.0 (260.79) | 142.5 (459.76) | 37.1 (138.82) | 41.7 (116.55)
  Week 48: number analyzed (Participants) | 190 | 197 | 83 | 77 | 40 | 48
  Week 48 | 59.6 (526.51) | 70.0 (366.63) | 18.8 (91.47) | 25.3 (108.19) | 42.5 (123.67) | 42.7 (148.11)
  Week 96: number analyzed (Participants) | 182 | 185 | 77 | 73 | 38 | 46
  Week 96 | 49.1 (245.14) | 56.1 (271.29) | 27.7 (204.80) | 13.3 (67.01) | 64.3 (183.16) | 22.3 (60.83)
  Week 144: number analyzed (Participants) | 155 | 160 | 66 | 59 | 31 | 41
  Week 144 | 44.1 (291.14) | 47.0 (169.68) | 18.8 (66.15) | 3.8 (25.03) | 42.6 (142.55) | 92.9 (397.69)
  Week 192: number analyzed (Participants) | 143 | 148 | 59 | 54 | 32 | 38
  Week 192 | 39.1 (217.89) | 54.5 (251.31) | 45.8 (156.88) | 19.9 (79.19) | 12.0 (40.56) | 55.1 (169.16)
  Week 240: number analyzed (Participants) | 134 | 133 | 55 | 52 | 28 | 34
  Week 240 | 96.8 (650.06) | 69.3 (374.67) | 21.7 (77.87) | 14.1 (45.22) | 17.5 (46.19) | 17.1 (48.41)
  Week 288: number analyzed (Participants) | 89 | 97 | 30 | 31 | 6 | 16
  Week 288 | 18.2 (93.28) | 53.1 (250.87) | 7.9 (30.09) | 230.2 (1092.11) | 0.0 (0.00) | 34.1 (102.87)

7. Secondary Outcome: Number of New or Newly Enlarging T2 Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The T2 lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
lesions
  Week 48: number analyzed (Participants) | 198 | 201 | 84 | 81 | 42 | 50
  Week 48 | 1.6 (4.07) | 2.2 (6.15) | 2.7 (4.96) | 2.4 (5.45) | 3.4 (6.57) | 2.1 (3.83)
  Week 96: number analyzed (Participants) | 191 | 192 | 78 | 77 | 40 | 47
  Week 96 | 3.4 (8.35) | 4.1 (10.01) | 3.8 (7.24) | 2.9 (6.78) | 4.9 (8.51) | 3.4 (5.13)
  Week 144: number analyzed (Participants) | 163 | 168 | 67 | 63 | 35 | 44
  Week 144 | 4.2 (9.81) | 5.2 (10.01) | 4.0 (7.27) | 4.3 (10.12) | 5.7 (9.45) | 5.2 (9.68)
  Week 192: number analyzed (Participants) | 151 | 155 | 61 | 56 | 33 | 40
  Week 192 | 5.8 (14.04) | 7.5 (15.14) | 5.6 (10.09) | 5.6 (14.19) | 5.5 (9.94) | 5.6 (13.35)
  Week 240: number analyzed (Participants) | 139 | 142 | 55 | 55 | 30 | 37
  Week 240 | 7.4 (17.09) | 9.5 (20.33) | 8.2 (14.87) | 7.7 (17.89) | 6.8 (11.74) | 7.5 (16.76)
  Week 288: number analyzed (Participants) | 123 | 123 | 45 | 49 | 26 | 32
  Week 288 | 8.2 (18.53) | 12.4 (28.23) | 7.5 (13.89) | 10.4 (22.05) | 8.9 (15.04) | 6.0 (8.90)

8. Secondary Outcome: Volume of New or Newly Enlarging T2 Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The T2 lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
mm^3
  Baseline: number analyzed (Participants) | 209 | 220 | 104 | 99 | 47 | 60
  Baseline | 10231.9 (11214.17) | 10408.3 (12166.80) | 8883.7 (8570.10) | 10806.3 (12060.05) | 12628.9 (11258.69) | 13044.4 (14608.50)
  Week 48: number analyzed (Participants) | 194 | 199 | 84 | 78 | 40 | 50
  Week 48 | 9951.9 (10750.15) | 9849.6 (10986.36) | 8992.1 (7952.13) | 10114.5 (10121.61) | 11160.7 (9565.55) | 12979.0 (14415.86)
  Week 96: number analyzed (Participants) | 187 | 190 | 78 | 74 | 38 | 47
  Week 96 | 10331.3 (11359.81) | 10434.0 (12201.38) | 8645.2 (7787.60) | 9985.7 (10715.73) | 11318.1 (9873.73) | 13974.1 (15432.10)
  Week 144: number analyzed (Participants) | 162 | 167 | 67 | 61 | 34 | 44
  Week 144 | 9930.1 (10686.26) | 10280.7 (11324.58) | 8829.4 (7482.93) | 9792.3 (9842.28) | 10188.5 (8064.09) | 12949.7 (14036.15)
  Week 192: number analyzed (Participants) | 149 | 154 | 61 | 55 | 32 | 40
  Week 192 | 9837.7 (10845.04) | 10760.0 (11987.16) | 9077.6 (7794.52) | 10576.3 (12029.26) | 10421.9 (8773.41) | 11671.5 (13124.47)
  Week 240: number analyzed (Participants) | 138 | 141 | 55 | 54 | 29 | 37
  Week 240 | 10611.2 (11633.95) | 11087.5 (12464.90) | 9711.1 (8709.46) | 10591.4 (11613.26) | 11009.9 (9551.94) | 12254.4 (13732.10)
  Week 288: number analyzed (Participants) | 121 | 122 | 45 | 49 | 26 | 32
  Week 288 | 9611.8 (9447.18) | 9800.8 (11279.84) | 8819.8 (8866.90) | 10537.6 (10684.47) | 11586.3 (9728.19) | 10404.8 (12245.75)

9. Secondary Outcome: Number of T1 Hypointense Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The T1 hypointense lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
lesions
  Week 48: number analyzed (Participants) | 183 | 184 | 79 | 76 | 41 | 48
  Week 48 | 0.8 (2.13) | 1.0 (2.37) | 1.8 (3.81) | 1.7 (3.71) | 2.0 (4.22) | 1.3 (2.64)
  Week 96: number analyzed (Participants) | 171 | 178 | 75 | 72 | 39 | 45
  Week 96 | 1.7 (3.63) | 1.9 (3.91) | 1.8 (3.33) | 2.1 (5.00) | 3.0 (5.85) | 1.9 (3.44)
  Week 144: number analyzed (Participants) | 148 | 155 | 63 | 53 | 32 | 41
  Week 144 | 2.0 (4.61) | 2.8 (5.19) | 2.0 (3.69) | 2.6 (7.02) | 3.1 (6.20) | 2.9 (5.19)
  Week 192: number analyzed (Participants) | 141 | 145 | 58 | 53 | 33 | 38
  Week 192 | 2.9 (7.03) | 3.4 (6.79) | 2.9 (5.12) | 3.8 (10.71) | 3.3 (6.74) | 3.0 (7.14)
  Week 240: number analyzed (Participants) | 134 | 136 | 55 | 53 | 29 | 34
  Week 240 | 3.4 (8.25) | 4.8 (9.39) | 4.0 (7.52) | 4.9 (13.30) | 4.0 (8.06) | 4.2 (10.20)
  Week 288: number analyzed (Participants) | 88 | 94 | 30 | 32 | 6 | 16
  Week 288 | 2.7 (5.72) | 5.9 (12.02) | 4.5 (7.38) | 3.6 (4.51) | 1.0 (1.10) | 5.6 (6.81)

10. Secondary Outcome: Volume of T1 Hypointense Lesions as Measured by Magnetic Resonance Imaging (MRI)
Description: The T1 hypointense lesions was evaluated using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
mm^3
  Baseline: number analyzed (Participants) | 209 | 220 | 104 | 99 | 47 | 60
  Baseline | 3640.1 (5598.31) | 3447.3 (4900.96) | 2754.2 (3552.30) | 3623.1 (5549.13) | 3204.3 (4221.55) | 3572.6 (4915.24)
  Week 48: number analyzed (Participants) | 190 | 197 | 83 | 77 | 40 | 48
  Week 48 | 3829.5 (5824.26) | 3715.5 (5112.21) | 2891.9 (3034.00) | 3936.0 (5271.89) | 3271.0 (4157.24) | 3743.3 (5374.24)
  Week 96: number analyzed (Participants) | 183 | 186 | 77 | 73 | 38 | 46
  Week 96 | 3841.2 (5682.74) | 3853.7 (5428.66) | 2921.0 (3327.93) | 3849.4 (5167.13) | 3510.4 (4672.80) | 3949.7 (5018.63)
  Week 144: number analyzed (Participants) | 157 | 164 | 67 | 58 | 33 | 42
  Week 144 | 3767.4 (4969.23) | 4074.0 (5413.85) | 3145.6 (3366.27) | 4006.9 (5062.08) | 3499.2 (4198.50) | 4126.1 (5695.44)
  Week 192: number analyzed (Participants) | 145 | 149 | 60 | 54 | 32 | 38
  Week 192 | 3834.9 (4942.19) | 4177.4 (5301.68) | 3385.4 (3575.44) | 4330.0 (5136.67) | 3592.0 (4069.39) | 4089.3 (4996.13)
  Week 240: number analyzed (Participants) | 135 | 137 | 55 | 52 | 28 | 34
  Week 240 | 4038.6 (5145.85) | 4238.2 (5248.84) | 3406.4 (3936.73) | 3823.9 (4274.82) | 3503.4 (3933.75) | 4057.7 (5223.62)
  Week 288: number analyzed (Participants) | 113 | 121 | 40 | 45 | 20 | 29
  Week 288 | 3603.3 (4394.60) | 3973.1 (5202.05) | 3350.6 (4140.34) | 4187.5 (4835.43) | 3264.9 (3639.91) | 2959.1 (3918.62)

11. Secondary Outcome: Percent Change From Baseline in Brain Atrophy
Description: Brain atrophy was measured using magnetic resonance imaging (MRI) technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
percent change
  Change at Week 48: number analyzed (Participants) | 162 | 162 | 56 | 64 | 33 | 42
  Change at Week 48 | -1.206 (1.1006) | -1.263 (1.0848) | -1.487 (1.3086) | -1.320 (1.4021) | -1.496 (1.1316) | -1.414 (1.1882)
  Change at Week 96: number analyzed (Participants) | 144 | 145 | 50 | 56 | 30 | 37
  Change at Week 96 | -1.372 (1.1382) | -1.500 (1.0893) | -1.589 (1.3630) | -1.775 (1.7191) | -1.883 (1.2383) | -1.810 (1.4556)
  Change at Week 144: number analyzed (Participants) | 122 | 133 | 44 | 49 | 28 | 36
  Change at Week 144 | -1.708 (1.4109) | -1.876 (1.2604) | -2.139 (1.5884) | -2.353 (1.7897) | -2.386 (1.3168) | -2.252 (2.2124)
  Change at Week 192: number analyzed (Participants) | 114 | 120 | 41 | 45 | 29 | 36
  Change at Week 192 | -2.138 (1.6831) | -2.117 (1.4000) | -2.230 (1.7755) | -2.476 (1.7062) | -2.645 (1.2284) | -2.417 (2.0486)
  Change at Week 240: number analyzed (Participants) | 92 | 95 | 37 | 40 | 18 | 26
  Change at Week 240 | -2.313 (1.6309) | -2.253 (1.3721) | -2.271 (1.4817) | -2.593 (1.9043) | -2.249 (1.2985) | -2.790 (2.2188)
  Change at Week 288: number analyzed (Participants) | 71 | 72 | 25 | 30 | 15 | 23
  Change at Week 288 | -2.216 (1.5744) | -2.271 (1.2193) | -2.470 (1.6757) | -2.849 (1.9648) | -2.657 (1.7051) | -2.496 (1.3699)

12. Secondary Outcome: Percent Change From Baseline in Magnetization Transfer Ratio (MTR)
Description: Magnetization Transfer Ratio (MTR) was measured using MRI technique.
Time Frame: Baseline up to Week 288
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 213 | 222 | 105 | 103 | 49 | 60
percent change
  Change at Week 48: number analyzed (Participants) | 126 | 118 | 49 | 56 | 20 | 23
  Change at Week 48 | -0.325 (5.4932) | -0.383 (4.8621) | 1.034 (7.3548) | -0.567 (4.4766) | -0.081 (13.6416) | -0.334 (1.5103)
  Change at Week 96: number analyzed (Participants) | 118 | 113 | 46 | 50 | 20 | 20
  Change at Week 96 | -0.427 (6.6493) | -0.532 (4.9880) | 1.630 (7.6584) | -0.947 (7.0771) | -4.269 (12.6065) | 0.215 (1.4270)
  Change at Week 144: number analyzed (Participants) | 103 | 107 | 45 | 37 | 19 | 24
  Change at Week 144 | -0.042 (9.2548) | 0.509 (7.2692) | 1.525 (8.6421) | 1.411 (12.2825) | -4.460 (10.3887) | 3.119 (8.1676)
  Change at Week 192: number analyzed (Participants) | 100 | 100 | 42 | 41 | 25 | 23
  Change at Week 192 | 1.038 (10.8680) | 0.955 (8.6105) | 3.012 (9.3831) | 3.103 (13.0046) | 1.384 (15.7611) | 3.841 (10.8600)
  Change at Week 240: number analyzed (Participants) | 91 | 90 | 40 | 42 | 23 | 20
  Change at Week 240 | -0.002 (15.6190) | 1.647 (8.3094) | 3.213 (9.6621) | 4.108 (13.8103) | 2.959 (16.8386) | 0.673 (25.9962)
  Change at Week 288: number analyzed (Participants) | 65 | 71 | 19 | 25 | 5 | 14
  Change at Week 288 | 0.002 (4.0206) | -0.391 (4.6415) | -0.666 (2.0741) | -0.622 (2.2922) | -0.466 (0.9410) | -1.114 (2.4539)

13. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36®) at Week 384
Description: The SF-36 is a brief (36-item) scale reflecting the impact of both dysfunctions and general health perception the questionnaire measures: 1.physical function (PF),2. role physical (RF),3. bodily pain (BP),4. role emotional (RE),5. social function (SF), 6. general health (GH),7. vitality (VT), 8. mental health (MH). Items 1-4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. The questions related to each dimension are scored on a scale from 0 (worst score) to 100 (best score), with higher scores indicating better function.
Time Frame: Baseline, Week 384
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
score on a scale
  Baseline: Physical Functioning Score: number analyzed (Participants) | 494 | 487 | 244 | 240 | 115 | 112
  Baseline: Physical Functioning Score | 68.48 (25.938) | 71.78 (24.849) | 69.67 (24.481) | 67.97 (26.279) | 69.10 (25.226) | 68.20 (25.370)
  Change at Week 384: Physical Functioning Score: number analyzed (Participants) | 236 | 215 | 90 | 97 | 43 | 48
  Change at Week 384: Physical Functioning Score | 0.73 (21.972) | -4.79 (24.641) | -7.37 (22.253) | -6.89 (23.194) | -6.19 (21.719) | -6.25 (28.350)
  Baseline: Role-Physical Score: number analyzed (Participants) | 494 | 486 | 244 | 238 | 114 | 112
  Baseline: Role-Physical Score | 56.46 (41.254) | 58.42 (41.280) | 56.35 (40.896) | 59.87 (41.747) | 55.26 (40.390) | 53.57 (42.029)
  Change at Week 384: Role-Physical Score: number analyzed (Participants) | 232 | 215 | 90 | 94 | 43 | 48
  Change at Week 384: Role-Physical Score | 3.20 (48.259) | -2.75 (47.283) | -10.00 (43.188) | -8.24 (53.177) | -12.21 (40.595) | -1.04 (54.568)
  Baseline: Bodily-Pain Score: number analyzed (Participants) | 494 | 490 | 244 | 240 | 115 | 112
  Baseline: Bodily-Pain Score | 69.68 (25.587) | 70.42 (24.688) | 68.51 (26.163) | 69.44 (26.016) | 69.30 (25.766) | 68.59 (26.102)
  Change at Week 384: Bodily-Pain Score: number analyzed (Participants) | 237 | 216 | 90 | 97 | 43 | 48
  Change at Week 384: Bodily-Pain Score | 1.32 (28.525) | -1.47 (25.779) | -2.92 (23.486) | -4.36 (25.935) | -3.60 (22.138) | -4.46 (33.297)
  Baseline: General Health Score: number analyzed (Participants) | 493 | 489 | 240 | 238 | 115 | 110
  Baseline: General Health Score | 53.99 (21.563) | 55.44 (20.768) | 54.45 (18.690) | 52.42 (20.028) | 51.21 (18.707) | 52.58 (19.675)
  Change at Week 384: General Health Score: number analyzed (Participants) | 234 | 213 | 86 | 95 | 42 | 47
  Change at Week 384: General Health Score | 0.87 (18.744) | -2.12 (20.595) | -2.28 (16.752) | -0.52 (22.035) | -5.64 (18.270) | 1.21 (21.674)
  Baseline: Vitality Score: number analyzed (Participants) | 492 | 486 | 242 | 239 | 115 | 111
  Baseline: Vitality Score | 50.48 (20.966) | 52.21 (19.842) | 50.63 (19.130) | 50.64 (21.069) | 51.30 (19.703) | 50.33 (20.019)
  Change at Week 384: Vitality Score: number analyzed (Participants) | 235 | 214 | 87 | 96 | 41 | 47
  Change at Week 384: Vitality Score | 1.11 (19.857) | -0.73 (19.033) | -4.67 (17.934) | 0.40 (20.822) | -6.71 (20.236) | 1.03 (19.829)
  Baseline: Social Functioning Score: number analyzed (Participants) | 494 | 490 | 244 | 239 | 115 | 112
  Baseline: Social Functioning Score | 71.46 (24.451) | 71.53 (24.394) | 69.67 (24.581) | 72.23 (24.699) | 69.02 (24.688) | 69.53 (25.100)
  Change at Week 384: Social Functioning Score: number analyzed (Participants) | 237 | 216 | 90 | 96 | 43 | 48
  Change at Week 384: Social Functioning Score | -2.16 (25.575) | -3.30 (24.912) | -5.69 (22.184) | -2.08 (27.724) | -10.76 (34.350) | -0.52 (25.780)
  Baseline: Role-Emotional Score: number analyzed (Participants) | 491 | 485 | 241 | 238 | 115 | 111
  Baseline: Role-Emotional Score | 64.87 (40.653) | 65.57 (40.015) | 62.86 (42.715) | 62.61 (41.280) | 60.29 (41.393) | 64.26 (41.854)
  Change at Week 384: Role-Emotional Score: number analyzed (Participants) | 233 | 214 | 90 | 96 | 43 | 47
  Change at Week 384: Role-Emotional Score | 0.43 (49.950) | 0.47 (43.513) | -12.22 (42.532) | 4.17 (44.656) | -13.18 (42.501) | -3.55 (48.769)
  Baseline: Mental Health Score: number analyzed (Participants) | 492 | 486 | 242 | 239 | 115 | 111
  Baseline: Mental Health Score | 65.01 (19.818) | 66.24 (19.060) | 65.42 (17.658) | 65.15 (19.233) | 62.30 (17.347) | 63.61 (18.414)
  Change at Week 384: Mental Health Score: number analyzed (Participants) | 235 | 214 | 87 | 96 | 41 | 47
  Change at Week 384: Mental Health Score | 1.32 (19.715) | 2.31 (18.095) | -3.91 (19.897) | 2.33 (17.524) | -0.29 (21.989) | -2.06 (20.066)
  Baseline: Mental Component Score: number analyzed (Participants) | 488 | 480 | 237 | 235 | 114 | 108
  Baseline: Mental Component Score | 45.40 (11.130) | 45.63 (10.272) | 45.13 (10.932) | 45.31 (10.907) | 44.00 (10.702) | 45.03 (10.642)
  Change at Week 384: Mental Component Score: number analyzed (Participants) | 226 | 211 | 85 | 92 | 41 | 45
  Change at Week 384: Mental Component Score | 0.05 (12.415) | 0.87 (10.028) | -2.55 (10.328) | 1.97 (10.657) | -2.59 (12.895) | 0.08 (10.328)
  Baseline: Physical Component Score: number analyzed (Participants) | 488 | 480 | 237 | 235 | 114 | 108
  Baseline: Physical Component Score | 43.53 (9.884) | 44.44 (10.048) | 43.74 (9.739) | 43.56 (10.267) | 43.68 (10.359) | 43.15 (10.091)
  Change at Week 384: Physical Component Score: number analyzed (Participants) | 226 | 211 | 85 | 92 | 41 | 45
  Change at Week 384: Physical Component Score | 0.55 (9.373) | -1.94 (10.532) | -2.29 (8.929) | -3.25 (9.998) | -2.70 (8.860) | -1.59 (10.765)

14. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions Questionnaire (EQ-5D) Health Survey - EQ-5D Index Score at Week 384
Description: The EQ-5D is a generic health-related quality of life instrument consisting of 2 components, EQ-5D index score and EQ-VAS. The EQ-5D provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to indicate whether he or she has (1) "no problems", (2) "some problems", or (3) "severe problems". A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 384
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
score on a scale
  Baseline: number analyzed (Participants) | 488 | 484 | 239 | 239 | 115 | 112
  Baseline | 0.73 (0.210) | 0.73 (0.222) | 0.72 (0.223) | 0.71 (0.244) | 0.71 (0.246) | 0.72 (0.189)
  Change at Week 384: number analyzed (Participants) | 230 | 212 | 86 | 96 | 42 | 48
  Change at Week 384 | 0.01 (0.251) | 0.00 (0.233) | -0.07 (0.269) | 0.00 (0.249) | -0.04 (0.253) | -0.03 (0.241)

15. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions Questionnaire (EQ-5D) Health Survey - Visual Analog Scale (VAS) at Week 384
Description: The EQ-5D is a generic health-related quality of life instrument consisting of 2 components, EQ-5D index score and EQ-VAS. In EQ-VAS participants are asked to rate their current health on a 20 centimeter (cm) scale from 0 to 100 where 0 represents "worst imaginable health state" and 100 represents "best imaginable health state". A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 384
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
score on a scale
  Baseline: number analyzed (Participants) | 492 | 488 | 243 | 238 | 113 | 112
  Baseline | 70.97 (18.460) | 70.48 (19.993) | 70.40 (17.630) | 69.44 (19.907) | 66.80 (18.846) | 69.07 (20.094)
  Change at Week 384: number analyzed (Participants) | 235 | 215 | 91 | 95 | 42 | 48
  Change at Week 384 | -0.48 (19.631) | -1.67 (18.855) | -7.24 (18.419) | -3.17 (22.003) | -1.71 (25.330) | -4.11 (16.270)

16. Secondary Outcome: Change From Baseline in Visual Function Test Scores at Week 384
Description: Participants were tested using the contrast level of 100%, 2.5%, and 1.25% charts, and the scores were defined as the number of letters identified correctly for each chart (the maximum score was 60). Higher scores indicate better functioning. A positive change from baseline indicates better functioning.
Time Frame: Baseline, Week 384
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BG00012 240 mg BID (Prior BG00012 240 mg BID) | BG00012 240 mg TID (Prior BG00012 240 mg TID) | BG00012 240 mg BID (Prior BG00012 Matched Placebo) | BG00012 240 mg TID (Prior BG00012 Matched Placebo) | BG00012 240 mg BID (Prior Glatiramer Acetate [GA]) | BG00012 240 mg TID (Prior Glatiramer Acetate [GA])
Number analyzed (Participants) | 501 | 502 | 249 | 248 | 118 | 118
score on a scale
  Baseline: 100% Chart | 54.7 (7.95) | 55.0 (7.84) | 55.1 (7.26) | 54.8 (7.12) | 54.3 (8.26) | 55.0 (6.73)
  Change at Week 384: 100% Chart: number analyzed (Participants) | 231 | 216 | 87 | 99 | 42 | 50
  Change at Week 384: 100% Chart | -0.4 (6.76) | -1.9 (6.81) | -1.4 (8.48) | -1.2 (7.53) | -1.6 (8.05) | -0.7 (5.17)
  Baseline: 2.5% Chart | 32.4 (12.17) | 32.6 (11.76) | 32.4 (11.42) | 32.3 (11.99) | 31.8 (12.36) | 31.7 (12.41)
  Change at Week 384: 2.5% Chart: number analyzed (Participants) | 231 | 216 | 87 | 99 | 42 | 50
  Change at Week 384: 2.5% Chart | -2.4 (10.77) | -3.3 (10.43) | -1.5 (11.77) | -4.9 (11.14) | -4.0 (11.90) | -2.1 (9.86)
  Baseline: 1.25% Chart: number analyzed (Participants) | 499 | 502 | 249 | 247 | 118 | 118
  Baseline: 1.25% Chart | 24.1 (12.45) | 24.2 (12.28) | 23.8 (12.11) | 23.7 (12.96) | 23.4 (11.76) | 22.2 (13.25)
  Change at Week 384: 1.25% Chart: number analyzed (Participants) | 231 | 216 | 87 | 99 | 42 | 50
  Change at Week 384: 1.25% Chart | -5.8 (13.39) | -6.0 (11.77) | -4.1 (13.04) | -7.4 (12.42) | -6.7 (13.78) | -5.0 (12.74)

ADVERSE EVENTS:
Time Frame: From start of the study up to follow-up (up to Week 561)
Description: Safety population included all participants who had any post-baseline safety follow-up in study NCT00835770, defined as any treatment emergent AE in Study NCT00835770 or any post-baseline laboratory, vital signs, or physical exam assessment in study NCT00835770, and received at least one dose of study treatment in study NCT00835770.
Arm/Group | BG00012 240 mg BID | BG00012 240 mg TID
All-Cause Mortality (participants affected / at risk) | 5/868 | 6/868
Serious Adverse Events (participants affected / at risk) | 279/868 | 272/868
Other Adverse Events (participants affected / at risk) | 779/868 | 767/868
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 240 mg BID (N=868) | BG00012 240 mg TID (N=868)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 5
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Wolff-parkinson-white syndrome (Cardiac disorders) | 1 | 0
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 | 1
Limb malformation (Congenital, familial and genetic disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 2 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal ischaemia (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Capsular contracture associated with breast implant (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Serositis (General disorders) | 0 | 1
Treatment failure (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 3 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 7
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 4
Bacterial infection (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Chronic sinusitis (Infections and infestations) | 0 | 2
Chronic tonsillitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 2 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 3
Infected skin ulcer (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Papilloma viral infection (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Peritonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (PML) (Infections and infestations) | 0 | 1
Pulmonary tuberculoma (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Scrub typhus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 10 | 4
Urosepsis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accident at work (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 13 | 18
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 4
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 3 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 5
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 5
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Investigation (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowenoid papulosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Complex partial seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 3 | 2
Dementia (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Multiple sclerosis (Nervous system disorders) | 4 | 2
Multiple sclerosis relapse (Nervous system disorders) | 116 | 122
Muscle spasticity (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 2
Optic neuritis (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 2 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Radiculitis (Nervous system disorders) | 1 | 0
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 2 | 1
Sciatica (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 2
Uhthoff's phenomenon (Nervous system disorders) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0
Catatonia (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 3
Drug abuse (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 2
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Morbid thoughts (Psychiatric disorders) | 1 | 0
Neurosis (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Psychotic behaviour (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Breast necrosis (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 2
Cystocele (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 3
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 1 | 3
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominoplasty (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0
Bladder neck suspension (Surgical and medical procedures) | 0 | 1
Bunion operation (Surgical and medical procedures) | 0 | 1
Caesarean section (Surgical and medical procedures) | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Cochlea implant (Surgical and medical procedures) | 0 | 1
Cystocele repair (Surgical and medical procedures) | 1 | 0
Female sterilisation (Surgical and medical procedures) | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Mammoplasty (Surgical and medical procedures) | 1 | 0
Medical device change (Surgical and medical procedures) | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1
Ovarian cystectomy (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 1 | 0
Postoperative care (Surgical and medical procedures) | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BG00012 240 mg BID (N=868) | BG00012 240 mg TID (N=868)
Lymphopenia (Blood and lymphatic system disorders) | 52 | 42
Abdominal pain (Gastrointestinal disorders) | 50 | 55
Abdominal pain upper (Gastrointestinal disorders) | 69 | 76
Diarrhoea (Gastrointestinal disorders) | 111 | 118
Nausea (Gastrointestinal disorders) | 56 | 61
Vomiting (Gastrointestinal disorders) | 42 | 45
Fatigue (General disorders) | 100 | 102
Pyrexia (General disorders) | 47 | 43
Bronchitis (Infections and infestations) | 82 | 98
Gastroenteritis (Infections and infestations) | 52 | 33
Herpes zoster (Infections and infestations) | 47 | 38
Influenza (Infections and infestations) | 87 | 67
Nasopharyngitis (Infections and infestations) | 220 | 226
Pharyngitis (Infections and infestations) | 44 | 50
Sinusitis (Infections and infestations) | 65 | 63
Upper respiratory tract infection (Infections and infestations) | 143 | 136
Urinary tract infection (Infections and infestations) | 196 | 164
Fall (Injury, poisoning and procedural complications) | 60 | 63
Alanine aminotransferase increased (Investigations) | 53 | 59
Albumin urine present (Investigations) | 66 | 62
Lymphocyte count decreased (Investigations) | 56 | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 97 | 115
Back pain (Musculoskeletal and connective tissue disorders) | 125 | 125
Muscle spasms (Musculoskeletal and connective tissue disorders) | 38 | 49
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 35 | 49
Pain in extremity (Musculoskeletal and connective tissue disorders) | 102 | 92
Dizziness (Nervous system disorders) | 60 | 45
Headache (Nervous system disorders) | 145 | 131
Hypoaesthesia (Nervous system disorders) | 64 | 49
Multiple sclerosis relapse (Nervous system disorders) | 324 | 335
Paraesthesia (Nervous system disorders) | 57 | 59
Anxiety (Psychiatric disorders) | 31 | 46
Depression (Psychiatric disorders) | 102 | 87
Insomnia (Psychiatric disorders) | 52 | 51
Haematuria (Renal and urinary disorders) | 49 | 61
Microalbuminuria (Renal and urinary disorders) | 55 | 61
Proteinuria (Renal and urinary disorders) | 76 | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 66
Erythema (Skin and subcutaneous tissue disorders) | 47 | 32
Pruritus (Skin and subcutaneous tissue disorders) | 50 | 38
Rash (Skin and subcutaneous tissue disorders) | 45 | 40
Flushing (Vascular disorders) | 170 | 165
Hot flush (Vascular disorders) | 44 | 53
Hypertension (Vascular disorders) | 51 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT00835770/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT00835770/SAP_001.pdf